CLINICAL TRIAL: NCT00286325
Title: Rituximab in the Treatment of Patients With Bullous Pemphigoid
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013763
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Results first posted 2012-10-22 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2012-09

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Rituximab (Experimental): Open label study all subjects treated with rituximab
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Infusion of 1000 mg of rituximab on day 0 and day 14
  Other Names: rituxan

SUMMARY:
This study will determine the safety of treatment of bullous pemphigoid in patients resistant to therapy with systemic corticosteroids, with rituximab plus systemic corticosteroids.

DETAILED DESCRIPTION:
Bullous pemphigoid (BP) is an autoimmune blistering disease characterized clinically by the presence of severely itchy, tense blisters located over the trunk and extremities. BP is the most common of the autoimmune blistering diseases with an incidence of approximately 10 per 1,000,000 population(1;2). In addition, BP occurs more frequently in the elderly. Routine histopathology reveals a sub-epidermal blister most often with large numbers of eosinophils. Direct immunofluorescence of the skin of patients with BP reveals a linear band of C3 and IgG at the basement membrane zone. Examination of the sera of patients shows the presence of a circulating anti-basement membrane zone autoantibody. This antibody has been found to be directed against a 180 kd protein of the basement membrane zone type XVII collagen (BPAg2) and against a 230 kd protein (BPAg1) found in the epidermal hemi-desmosome(3;4).

BP is a severe disease most often requiring therapy with high dose systemic corticosteroids (0.75 - 1.0 mg/kg/day) often for months(5). In addition, relapses are common and the additional use of immunosuppressive drugs such as azathioprine, methotrexate, cyclosporine A and others are needed to minimize the dose of systemic corticosteroids. The 1-year mortality of BP has been estimated to range from 10 - 30%(1;6). Currently treatment of patients with BP consists of initial use of systemic corticosteroids (0.75 - 1.0 mg/kg/day). Control of symptoms and new blister formation is most often achieved within 1 month and systemic corticosteroids are then tapered. As many as 33 - 50% of patients may not be able to be tapered to clinically acceptable levels of systemic corticosteroids, requiring the addition of systemic immunosuppression often with azathioprine. Approximately 66% of patients require long term treatment with immunosuppressive medication to maintain control of their blistering.(5;7;8) The need for long term systemic corticosteroid therapy often with systemic immunosuppression in an elderly population results in a significant morbidity and mortality in patients with BP. New therapeutic interventions that would potentially allow for the more rapid discontinuation of prednisone, avoidance of systemic immuno- suppression and perhaps earlier clinical relapse would be of substantial benefit to patients with BP. The clinical and laboratory data has demonstrated that BP is an autoantibody mediated blistering disease. Taken together these observations suggest that the use of anti-CD20 antibody (Rituxan) may be useful in the treatment of patients with BP. We have previously treated a patient with BP and graft versus host disease with anti-CD20 and anti-CD25 and were able to achieve clinical and serological remission within 4 weeks of initiation of therapy(9). In addition, others and we have successfully utilized Rituxan for the treatment of pemphigus vulgaris, another autoantibody mediated, autoimmune blistering disease(10-15)

ELIGIBILITY:
Inclusion Criteria:

* Patients with autoimmune blistering skin diseases with clinical, histologic and immunological criteria confirming the diagnosis of bullous pemphigoid
* Ongoing disease activity on 17.5 mg/day of prednisone or more

Exclusion Criteria:

* Current use of other immunosuppressive therapy such as azathioprine, cytoxan or mycophenolate mofetil within the last 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Hall, III, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Anolik JH, Campbell D, Felgar RE, Young F, Sanz I, Rosenblatt J, Looney RJ. The relationship of FcgammaRIIIa genotype to degree of B cell depletion by rituximab in the treatment of systemic lupus erythematosus. Arthritis Rheum. 2003 Feb;48(2):455-9. doi: 10.1002/art.10764. PMID 12571855
- [Background] Gupta N, Kavuru S, Patel D, Janson D, Driscoll N, Ahmed S, Rai KR. Rituximab-based chemotherapy for steroid-refractory autoimmune hemolytic anemia of chronic lymphocytic leukemia. Leukemia. 2002 Oct;16(10):2092-5. doi: 10.1038/sj.leu.2402676. PMID 12357362
- [Background] Leandro MJ, Edwards JC, Cambridge G. Clinical outcome in 22 patients with rheumatoid arthritis treated with B lymphocyte depletion. Ann Rheum Dis. 2002 Oct;61(10):883-8. doi: 10.1136/ard.61.10.883. PMID 12228157
- [Background] Maloney DG, Grillo-Lopez AJ, Bodkin DJ, White CA, Liles TM, Royston I, Varns C, Rosenberg J, Levy R. IDEC-C2B8: results of a phase I multiple-dose trial in patients with relapsed non-Hodgkin's lymphoma. J Clin Oncol. 1997 Oct;15(10):3266-74. doi: 10.1200/JCO.1997.15.10.3266. PMID 9336364
- [Background] McLaughlin P, Grillo-Lopez AJ, Link BK, Levy R, Czuczman MS, Williams ME, Heyman MR, Bence-Bruckler I, White CA, Cabanillas F, Jain V, Ho AD, Lister J, Wey K, Shen D, Dallaire BK. Rituximab chimeric anti-CD20 monoclonal antibody therapy for relapsed indolent lymphoma: half of patients respond to a four-dose treatment program. J Clin Oncol. 1998 Aug;16(8):2825-33. doi: 10.1200/JCO.1998.16.8.2825. PMID 9704735
- [Background] Pestronk A, Florence J, Miller T, Choksi R, Al-Lozi MT, Levine TD. Treatment of IgM antibody associated polyneuropathies using rituximab. J Neurol Neurosurg Psychiatry. 2003 Apr;74(4):485-9. doi: 10.1136/jnnp.74.4.485. PMID 12640069
- [Background] Piro LD, White CA, Grillo-Lopez AJ, Janakiraman N, Saven A, Beck TM, Varns C, Shuey S, Czuczman M, Lynch JW, Kolitz JE, Jain V. Extended Rituximab (anti-CD20 monoclonal antibody) therapy for relapsed or refractory low-grade or follicular non-Hodgkin's lymphoma. Ann Oncol. 1999 Jun;10(6):655-61. doi: 10.1023/a:1008389119525. PMID 10442187
- [Background] Reff ME, Carner K, Chambers KS, Chinn PC, Leonard JE, Raab R, Newman RA, Hanna N, Anderson DR. Depletion of B cells in vivo by a chimeric mouse human monoclonal antibody to CD20. Blood. 1994 Jan 15;83(2):435-45. PMID 7506951
- [Background] Stasi R, Pagano A, Stipa E, Amadori S. Rituximab chimeric anti-CD20 monoclonal antibody treatment for adults with chronic idiopathic thrombocytopenic purpura. Blood. 2001 Aug 15;98(4):952-7. doi: 10.1182/blood.v98.4.952. PMID 11493438
- [Background] Stasi R, Stipa E, Forte V, Meo P, Amadori S. Variable patterns of response to rituximab treatment in adults with chronic idiopathic thrombocytopenic purpura. Blood. 2002 May 15;99(10):3872-3. doi: 10.1182/blood-2002-02-0392. No abstract available. PMID 12014370
- [Background] Zaja F, Iacona I, Masolini P, Russo D, Sperotto A, Prosdocimo S, Patriarca F, de Vita S, Regazzi M, Baccarani M, Fanin R. B-cell depletion with rituximab as treatment for immune hemolytic anemia and chronic thrombocytopenia. Haematologica. 2002 Feb;87(2):189-95. PMID 11836170
- [Background] Bernard P, Bedane C, Bonnetblanc JM. Anti-BP180 autoantibodies as a marker of poor prognosis in bullous pemphigoid: a cohort analysis of 94 elderly patients. Br J Dermatol. 1997 May;136(5):694-8. PMID 9205501
- [Background] Cooper HL, Healy E, Theaker JM, Friedmann PS. Treatment of resistant pemphigus vulgaris with an anti-CD20 monoclonal antibody (Rituximab). Clin Exp Dermatol. 2003 Jul;28(4):366-8. doi: 10.1046/j.1365-2230.2003.01283.x. PMID 12823293
- [Background] Diaz LA, Ratrie H 3rd, Saunders WS, Futamura S, Squiquera HL, Anhalt GJ, Giudice GJ. Isolation of a human epidermal cDNA corresponding to the 180-kD autoantigen recognized by bullous pemphigoid and herpes gestationis sera. Immunolocalization of this protein to the hemidesmosome. J Clin Invest. 1990 Oct;86(4):1088-94. doi: 10.1172/JCI114812. PMID 1698819
- [Background] Dupuy A, Viguier M, Bedane C, Cordoliani F, Blaise S, Aucouturier F, Bonnetblanc JM, Morel P, Dubertret L, Bachelez H. Treatment of refractory pemphigus vulgaris with rituximab (anti-CD20 monoclonal antibody). Arch Dermatol. 2004 Jan;140(1):91-6. doi: 10.1001/archderm.140.1.91. PMID 14732665
- [Background] Giudice GJ, Liu Z, Diaz LA. An animal model of bullous pemphigoid: what can it teach us? Proc Assoc Am Physicians. 1995 Jul;107(2):237-41. PMID 8624858
- [Background] Goebeler M, Herzog S, Brocker EB, Zillikens D. Rapid response of treatment-resistant pemphigus foliaceus to the anti-CD20 antibody rituximab. Br J Dermatol. 2003 Oct;149(4):899-901. doi: 10.1046/j.1365-2133.2003.05580.x. No abstract available. PMID 14616397
- [Background] Herrmann G, Hunzelmann N, Engert A. Treatment of pemphigus vulgaris with anti-CD20 monoclonal antibody (rituximab). Br J Dermatol. 2003 Mar;148(3):602-3. doi: 10.1046/j.1365-2133.2003.05209_10.x. No abstract available. PMID 12653767
- [Background] Khumalo NP, Murrell DF, Wojnarowska F, Kirtschig G. A systematic review of treatments for bullous pemphigoid. Arch Dermatol. 2002 Mar;138(3):385-9. doi: 10.1001/archderm.138.3.385. PMID 11902990
- [Background] Korman NJ. Bullous pemphigoid. The latest in diagnosis, prognosis, and therapy. Arch Dermatol. 1998 Sep;134(9):1137-41. doi: 10.1001/archderm.134.9.1137. No abstract available. PMID 9762028
- [Background] Liu Z, Diaz LA, Troy JL, Taylor AF, Emery DJ, Fairley JA, Giudice GJ. A passive transfer model of the organ-specific autoimmune disease, bullous pemphigoid, using antibodies generated against the hemidesmosomal antigen, BP180. J Clin Invest. 1993 Nov;92(5):2480-8. doi: 10.1172/JCI116856. PMID 7693763
- [Background] Nousari HC, Anhalt GJ. Pemphigus and bullous pemphigoid. Lancet. 1999 Aug 21;354(9179):667-72. doi: 10.1016/S0140-6736(99)03007-X. PMID 10466686
- [Background] Roujeau JC, Lok C, Bastuji-Garin S, Mhalla S, Enginger V, Bernard P. High risk of death in elderly patients with extensive bullous pemphigoid. Arch Dermatol. 1998 Apr;134(4):465-9. doi: 10.1001/archderm.134.4.465. PMID 9554299
- [Background] Rzany B, Partscht K, Jung M, Kippes W, Mecking D, Baima B, Prudlo C, Pawelczyk B, Messmer EM, Schuhmann M, Sinkgraven R, Buchner L, Budinger L, Pfeiffer C, Sticherling M, Hertl M, Kaiser HW, Meurer M, Zillikens D, Messer G. Risk factors for lethal outcome in patients with bullous pemphigoid: low serum albumin level, high dosage of glucocorticosteroids, and old age. Arch Dermatol. 2002 Jul;138(7):903-8. doi: 10.1001/archderm.138.7.903. PMID 12071817
- [Background] Salopek TG, Logsetty S, Tredget EE. Anti-CD20 chimeric monoclonal antibody (rituximab) for the treatment of recalcitrant, life-threatening pemphigus vulgaris with implications in the pathogenesis of the disorder. J Am Acad Dermatol. 2002 Nov;47(5):785-8. doi: 10.1067/mjd.2002.126273. PMID 12399777
- [Background] Stanley JR, Hawley-Nelson P, Yuspa SH, Shevach EM, Katz SI. Characterization of bullous pemphigoid antigen: a unique basement membrane protein of stratified squamous epithelia. Cell. 1981 Jun;24(3):897-903. doi: 10.1016/0092-8674(81)90115-x. No abstract available. PMID 7018697
- [Background] Szabolcs P, Reese M, Yancey KB, Hall RP, Kurtzberg J. Combination treatment of bullous pemphigoid with anti-CD20 and anti-CD25 antibodies in a patient with chronic graft-versus-host disease. Bone Marrow Transplant. 2002 Sep;30(5):327-9. doi: 10.1038/sj.bmt.1703654. PMID 12209356
- [Background] Venning VA, Wojnarowska F. Lack of predictive factors for the clinical course of bullous pemphigoid. J Am Acad Dermatol. 1992 Apr;26(4):585-9. doi: 10.1016/0190-9622(92)70085-t. PMID 1597545
- [Background] Gault MH, Purchase L. Would decreased aluminum ingestion reduce the incidence of Alzheimer's disease? CMAJ. 1992 Sep 15;147(6):845-7. No abstract available. PMID 1285757
- [Background] Wojnarowska F, Kirtschig G, Highet AS, Venning VA, Khumalo NP; British Association of Dermatologists. Guidelines for the management of bullous pemphigoid. Br J Dermatol. 2002 Aug;147(2):214-21. doi: 10.1046/j.1365-2133.2002.04835.x. PMID 12174090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with bullous pemphigoid were recruited in dermatology clinics from 2005 - 2009.
Pre-assignment Details: Patient were screened for appropriate diagnosis, disease activity, prednisone dosage before entry into the study
Groups:
- Treated: Open label study subjects all treated with rituximab
Period: Overall Study
Arm/Group | Treated
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treated
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Secondary Outcome: Number of Days to Cessation of New Blister
Description: The first study visit in which patient reported and was confirmed to have no new blister or lesion formation .
Time Frame: 1 year
Population: Excluded subject with diagnosis of epidermolysis bullosa acquisita , made after study entry.
Measure: Median (Full Range); unit: Days
Arm/Group | Treated
Number analyzed (Participants) | 7
Days | 57 [13 to 163]

2. Primary Outcome: Primary Safety Endpoint
Description: The primary safety endpoint is the occurrence of treatment emergent adverse events including infections, infusion reactions and disease progression. These were determined by clinical evaluation and laboratory questions. Disease progression is defined as development of new blisters despite therapy. These are reported as the number of participants with a study related SAE.
Time Frame: 1 year
Population: The safety analysis was performed on all subjects
Measure: Number; unit: participants
Arm/Group | Treated
Number analyzed (Participants) | 8
participants
  Treatment emergent adverse events | 0
  Infusion reactions | 0
  Disease Progression | 1

3. Secondary Outcome: Systemic Corticosteroid Dose of 25% of Starting Dose or 10 mg/Day by Week 24
Description: Subject systemic corticosteroid dosage at week 24 was 25% of starting dose or 10 mg/day of prednisone or less
Time Frame: 24 weeks
Population: Excluded subject with epidermolysis bullosa acquisita diagnosed after study entry.
Measure: Number; unit: participants
Arm/Group | Treated
Number analyzed (Participants) | 7
participants | 7

4. Secondary Outcome: IgG Anti Bullous Pemphigoid (BP) 180 Measured in Units by ELISA at Week 24.
Description: IgG antibodies against BP 180 measured in units (by ELISA) for each participant at week 0 compared to value at week 24,
Time Frame: Week 0 and at 24 weeks
Population: Excluded subject with diagnosis of epidermolysis bullosa acquisita made after study entry, excluded one subject with no circulating antibodies measured at either time point.
Measure: Median (Full Range); unit: Elisa Units
Arm/Group | Treated
Number analyzed (Participants) | 6
Elisa Units | 40.5 [6 to 72]
Statistical Analysis 1: Comparison: Treated; Wilcoxon comparing week zero antibody value in units to week 24 antibody value in units; Test type: Superiority or Other; p = 0.0156, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: B Cell Number at Week 24
Description: Peripheral blood B cell number at week 24 compared to B cell number at week 0
Time Frame: Week 0 and at 24 weeks
Population: excluded subject with epidermolysis bullosa acquisita diagnosed after study entry
Measure: Median (Full Range); unit: B cells per microliter
Arm/Group | Treated
Number analyzed (Participants) | 7
B cells per microliter | 3.99 [1.41 to 137.6]
Statistical Analysis 1: Comparison: Treated; Comparison of B cell number at week 0 to b cell number in participants at week 24; Test type: Superiority or Other; p = 0.0078, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events related or possibly related to study drug
Arm/Group | Treated
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
Open label trial of rituximab in the treatment of 7 patients with the autoimmune blistering disease bullous pemphigoid.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No